CLINICAL TRIAL: NCT03889457
Title: Patients' Choice in Terms of Anticoagulant Therapy in Venous Thrombo- Embolism Disease. AntiCoagChoice Study
Brief Title: What Treatment for Patients With Phlebitis or Pulmonary Embolism ?
Acronym: AntiCoagChoice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Collaborators: SFMV (French Society of Vascular Medicine) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3002_AntiCoagChoice
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-02

CONDITIONS: Venous Thrombosis or Pulmonary Embolism
Keywords: Deep Vein Thrombosis; Superficial Vein Thrombosis; Anticoagulant; Patient Compliance; Preference; Venous Thrombosis; pulmonary embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with venous thromboembolic disease: Patients with deep vein thrombosis, superficial or muscular vein thrombosis, pulmonary embolism, over 18 years of age.
  Interventions: Other: anticoagulation choice

INTERVENTIONS:
Other: anticoagulation choice — Type of anticoagulant chosen by the patient (oral or injectable).

SUMMARY:
The objective of the "anticoagchoice" study is to analyze the preferences of people suffering from phlebitis, in terms of anticoagulant, to improve adherence to these treatments, to adapt the medical prescriptions.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is the third leading cause of cardiovascular death, with an increase in annual incidence with age. With the advent of direct oral anticoagulants, the management of deep vein thrombosis and pulmonary embolism has evolved in recent years and these treatments are widely prescribed. There are studies comparing the different anticoagulant treatments used in venous thrombosis, which show no inferiority of treatment (injectable or oral) compared to others. Drug delivery modalities have been shown to affect adherence, and thus treatment efficacy. It seems fundamental to focus on patients' drug preferences in VTE to ensure the best possible compliance. These preferences seem to depend on the personal history of each patient. In addition, no studies have been conducted on patient preferences for anticoagulant therapy for VTE: this is the goal of the "anticoagchoice" study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with deep vein thrombosis, superficial vein thrombosis, muscle vein thrombosis or pulmonary embolism, over 18 years of age.

No Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with deep vein thrombosis, superficial vein thrombosis, muscle vein thrombosis or pulmonary embolism, over 18 years of age in France (via the vascular doctors of the French Society of Vascular Médicine).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-02-12 (Estimated); Study Completion 2021-02-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to analyze patient treatment preferences in venous thromboembolic disease. | the time required for a consultation: 30 minutes
  The primary outcome: To compare the proportion of patients choosing oral anticoagulation vs patients choosing injectable route.

SECONDARY OUTCOMES:
compare patients choosing oral anticoagulation vs patients choosing an injectable route | the time required for a consultation: 30 minutes
  proportions of patients choosing an oral anticoagulation vs. patients choosing an injectable pathway depending on the duration of treatment (3 months, 6 months or more),
compare patients choosing oral anticoagulation vs patients choosing an injectable route | the time required for a consultation: 30 minutes
  Identify factors influencing these choices, depending on the characteristics of the patient (history, age, gender, social environment, personal experience).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mahe, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laneelle D, Le Brun C, Mauger C, Guillaumat J, Le Pabic E, Omarjee L, Mahe G; SFMV VTE Study Group. Patient Characteristics and Preferences Regarding Anticoagulant Treatment in Venous Thromboembolic Disease. Front Cardiovasc Med. 2021 Jun 21;8:675969. doi: 10.3389/fcvm.2021.675969. eCollection 2021. PMID 34235186